CLINICAL TRIAL: NCT04383353
Title: Burning Rock Pan-canceR Early DetectIon projeCT (PREDICT): a Prospective, Multicenter Study to Develop and Validate the Performance of a cfDNA Methylation Based Model on Early Cancer Detection
Brief Title: Pan-canceR Early DetectIon projeCT
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RSCD2020001
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Cancer
Keywords: cancer; cell-free DNA (cfDNA) methylation; early detection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer arm: Participants with new diagnosis of cancer, from whom a blood sample and contemporaneous tissue samples will be collected.
- Benign disease arm: Participants with benign diseases corresponding to the tumor types in the cancer arm, from whom a blood sample and contemporaneous tissue samples will be collected.
- Non-tumor arm (Healthy): Participants with no known presence of malignancies or benign diseases, from whom a blood sample will be collected.

SUMMARY:
PREDICT is a prospective, multi-center study for the early detection of pan-cancer through cell-free DNA (cfDNA) methylation based model, in which approximately 14,000 participants will be enrolled. The development and validation of the model will be conducted in participants with early stage cancers or benign diseases, along with non-tumor (healthy) individuals through a two-stage approach. The sensitivity and specificity of the model in cancer early detection will be evaluated, and the accuracy of the identification for tissue of origin will be obtained.

ELIGIBILITY:
Inclusion Criteria for Cancer Arm Participants:

* Able to provide a written informed consent.
* Able to provide sufficient and qualified blood samples for study tests.
* No prior or undergoing cancer treatment (local or systematic) with either of the following:
* A. Pathologically confirmed cancer diagnosis within 30 (±7) days prior to the study blood draw.
* B. High suspicious for cancer diagnosis by radiological or other routine clinical assessments, with confirmed cancer diagnosis through biopsy or surgical resection within 36 (±7) days after study blood draw.

Exclusion Criteria for Cancer Arm Participants:

* Insufficient qualified blood sample for study test.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 30 days prior to study blood draw.
* With other known malignant tumors or multiple primary tumors.

Inclusion Criteria for Benign Disease Arm Participants:

* Able to provide a written informed consent.
* Able to provide sufficient and qualified blood samples for study tests.
* Have either of the following:
* A. Pathological confirmed diagnosis of benign diseases within 90 (±7) days prior to the study blood draw, with no prior treatment such as surgical resection.
* B. High suspicious for benign diseases diagnosis by radiological or other routine clinical assessments, with confirmed benign diseases diagnosis within 36 (±7) days after study blood draw.

Exclusion Criteria for Benign Disease Arm Participants:

* Insufficient qualified blood sample for study test.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 30 days prior to study blood draw.

Inclusion Criteria for Non-Tumor Arm Participants:

* Able to provide a written informed consent.
* Able to provide sufficient and qualified blood samples for study tests.
* No cancer related symptoms within 30 days prior to study screening.
* Cancer history with curative treatment completed over 3 years without recurrence prior to study enrollment.

Exclusion Criteria for Non-Tumor Arm Participants:

* Insufficient qualified blood sample for study test.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 30 days prior to study blood draw.
* Recipient of anti-infectious therapy within 14 days prior to study blood draw.
* Have received or are undergoing curative cancer treatment within three years prior to study screening.
* With autoimmune or other diseases with severe comorbidities.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and assigned into three arms, including participants with new diagnosis of malignancy or corresponding benign disease, and participants without the presence of malignant or benign diseases.
Sampling Method: Non-Probability Sample
Enrollment: 14026 (Estimated)
Dates: Start 2020-07-21 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The cfDNA methylations profiles of patients with malignancies or benign diseases using pre-treatment biospecimens. | 32 months
The sensitivity and specificity of multi-cancer early detection and the accuracy of TOO identification via cfDNA methylation based model. | 32 months

SECONDARY OUTCOMES:
The sensitivity and specificity of cancer early detection and the accuracy of TOO identification via cfDNA methylation based model in pre-specified subgroups. | 32 months
The sensitivity and specificity of cancer early detection and the accuracy of TOO identification via cfDNA methylation based model in combination with clinicopathological characteristics or other biomarkers. | 32 months
The examinations related to cancer diagnosis from the participants who were identified as positive cases by cfDNA methylation based model while as healthy individuals by routine medical examinations. | 32 months
The sensitivity and specificity of cancer early detection and the accuracy of TOO identification via cfDNA methylation based model in the independent training and validation sets. | 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Hao Liu, M.D, Study Director — Guangzhou Burning Rock Dx Co., Ltd.
Locations (3):
- China (3):
  - Cancer Hospital, Chinese Academy of Medical Sciences & China National Cancer Center, Beijing, Beijing Municipality
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo B, Ma F, Liu H, Hu J, Rao L, Liu C, Jiang Y, Kuangzeng S, Lin X, Wang C, Lei Y, Si Z, Chen G, Zhou N, Liang C, Jiang F, Liu F, Dai W, Liu W, Gao Y, Li Z, Li X, Zhou G, Li B, Zhang Z, Nian W, Luo L, Liu X. Cell-free DNA methylation markers for differential diagnosis of hepatocellular carcinoma. BMC Med. 2022 Jan 14;20(1):8. doi: 10.1186/s12916-021-02201-3. PMID 35027051